CLINICAL TRIAL: NCT01110785
Title: Safety and Efficacy of the Addition of Simvastatin to Panitumumab in K-ras Mutant Advanced or Metastatic Colorectal Cancer Patients. A Single-Arm, Multicenter, Phase II Study Using a Simon Two Stage Design.
Brief Title: Simvastatin and Panitumumab in Treating Patients With Advanced or Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000671002; DUT-LUMC-30012009; EUDRACT-2009-014452-30; EU-21033; DUT-LUMC-RASTAT-P; NL-29611-058-09
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2011-04

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Panitumumab; Simvastatin

INTERVENTIONS:
Biological: panitumumab
Drug: simvastatin
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Simvastatin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving simvastatin together with panitumumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well simvastatin given together with panitumumab works in treating patients with advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if the proportion (at least 40%) of patients with K-ras mutant-type advanced or metastatic colorectal cancer are free from progression and alive based on RECIST criteria version 1.1 at 11 weeks after the first administration of panitumumab (i.e., 12.5 weeks after the scan at baseline at start of simvastatin).
* To determine if these results are comparable with historical results of k-ras wild-type colorectal carcinoma patients treated with panitumumab.
* To evaluate clinical signs of progression (according to RECIST criteria) in patients treated with this regimen.

Secondary

* To evaluate the safety of this regimen in these patients who have failed prior treatment with fluorouracil-, oxaliplatin-, and irinotecan-containing regimens.
* To evaluate the overall survival of patients who are treated with this regimen and have failed prior fluorouracil-, oxaliplatin-, and irinotecan-containing regimens.
* To evaluate the progression-free survival (based on RECIST criteria version 1.1) of these patients.
* To evaluate the objective response rate (based on RECIST criteria version 1.1) in these patients.
* To evaluate the correlation between skin toxicity and anti-tumor response in these patients.

Tertiary (exploratory)

* To evaluate the role of serum cholesterol as a biomarker during treatment with panitumumab and simvastatin.
* To correlate levels of serum cholesterol with treatment response and other factors, until progression of disease occurs.
* To investigate whether PTEN, PIK3CA, b-raf, ERK, and MEK status correlate with response to panitumumab in these patients.
* To investigate the role of single nucleotide polymorphisms related to the efficacy and metabolism of panitumumab as a predictor for response to panitumumab.
* To investigate the role of proteomics (e.g., EGF) as potential predictive markers for response to panitumumab and as potential biomarkers during treatment with panitumumab.

OUTLINE: This is a multicenter study.

Patients receive oral simvastatin once daily on days 1-14 and panitumumab IV over 30-90 minutes on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for biomarker and other analyses.

After completion of study treatment, patients are followed for 30 days and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer

  * Advanced or metastatic disease
* Failed prior fluorouracil-, oxaliplatin- and irinotecan-containing regimens

  * In case of progressive disease within 6 months after start of adjuvant fluorouracil-, oxaliplatin-, and irinotecan-containing regimens, the adjuvant therapy is considered to be treatment for metastatic disease
* Mutant-type k-ras status (mutation in codon 12, 13, or 61) on tumor material
* Measurable disease according to RECIST criteria version 1.1
* Progressive disease in the past 3 months according to RECIST criteria version 1.1
* No symptomatic brain metastases, defined as any symptoms during the past 6 months

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* WBC ≥ 2.0 x 10^9/L
* ANC ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 9 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 3 times ULN (≤ 5 times ULN in case of liver metastases)
* Creatinine clearance ≥ 60 mL/min
* Magnesium normal
* Calcium normal
* Creatine phosphokinase ≤ 2.5 times ULN
* Not pregnant or nursing
* Not planning to become pregnant within 6 months after the end of study treatment
* Fertile patients must use highly effective contraception during and for 6 months after completion of study therapy
* No noncompliance in previous studies
* No alcohol use > 4 units/day or unwilling to abstain from use
* No history of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or signs of interstitial lung disease on baseline CT scan
* No clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, or serious uncontrolled cardiac arrhythmia) < 1 year prior to study
* No symptomatic hypothyroidism
* No history of toxicity during statin use

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior EGFr-therapy, including monoclonal antibodies (e.g., panitumumab or cetuximab)
* No concurrent verapamil, amiodarone, or dronedarone or unwilling to abstain from use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients free from progression and alive at 11 weeks after the first dose of panitumumab measured by RECIST v 1.1

SECONDARY OUTCOMES:
Toxicity measured by NCICTC v 3.0
Median and mean overall survival
Median and mean progression-free survival
Objective response rate
Correlation between skin toxicity and response to treatment
Serum cholesterol and subsequent treatment response
Correlation between PTEN, PIK3CA, b-raf, ERK, and MEK status and objective response rate
Correlation between single nucleotide polymorphisms and objective response rate
Correlation between proteomics and objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gelderblom, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (4):
- Netherlands (4):
  - Reinier de Graaf Group - Delft, Delft
  - Leiden University Medical Center, Leiden
  - Diaconessenhuis Leiden, Leiden
  - HagaZiekenhuis - Locatie Leyenburg, The Hague